CLINICAL TRIAL: NCT04283136
Title: An Open-Label, Randomized, Single-Dose, 2-Part Crossover Study in Healthy Study Participants to Evaluate the Relative Bioavailability of 4 Padsevonil Product Variants and the Effect of Food on Padsevonil
Brief Title: A Study to Test the Blood Concentration of 4 Padsevonil Product Variants and the Effect of Food on Padsevonil
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizures
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP0081
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Healthy Participants; Epilepsy
Keywords: Phase 1; Padsevonil; Bioavailability; Food effect
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: In Part 1 a single oral dose of padsevonil 200 mg for the 4 different product variants and the padsevonil reference tablet will be administered to all subjects in the fasted state in a randomized 5-way crossover design. In order to explore the food interaction with padsevonil, in Part 2 a single oral dose of a padsevonil reference tablet at dose levels of 200 mg and 400 mg (2x 200mg tablets) will be administered to all subjects in the fasted and fed state in a randomized 4-way crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Type 1 tablet - part 1 (Active Comparator): Subjects will receive a single dose of padsevonil Type 1 tablet in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 1 Tablet 200 mg
- Type 2 tablet - part 1 (Experimental): Subjects will receive a single dose of padsevonil Type 2 tablet in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 2 Tablet
- Type 3 tablet - part 1 (Experimental): Subjects will receive a single dose of padsevonil Type 3 tablet in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 3 Tablet
- Type 4 tablet - part 1 (Experimental): Subjects will receive a single dose of padsevonil Type 4 tablet in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 4 Tablet
- Type 5 tablet - part 1 (Experimental): Subjects will receive a single dose of padsevonil Type 5 tablet in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 5 Tablet
- Type 1 tablet - part 2 (2 x 200 mg fasted) (Active Comparator): Subjects will receive a single 2 x 200 mg dose of padsevonil Type 1 tablet under fasting conditions in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 1 Tablet 200 mg
- Type 1 tablet - part 2 (2 x 200 mg fed) (Active Comparator): Subjects will receive a single 2 x 200 mg dose of padsevonil Type 1 tablet under fed conditions in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 1 Tablet 200 mg
- Type 1 tablet - part 2 (200 mg fasted) (Active Comparator): Subjects will receive a single 200 mg dose of padsevonil Type 1 tablet under fasting conditions in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 1 Tablet 200 mg
- Type 1 tablet - part 2 (200 mg fed) (Active Comparator): Subjects will receive a single 200 mg dose of padsevonil Type 1 tablet under fed conditions in the period defined by the pre-specified sequence they were randomized on to.
  Interventions: Drug: Padsevonil type 1 Tablet 200 mg

INTERVENTIONS:
Drug: Padsevonil type 1 Tablet 200 mg — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Subjects will receive a padsevonil type 1 tablet in a pre-specified sequence during the Treatment Period.
  Arms: Type 1 tablet - part 1; Type 1 tablet - part 2 (2 x 200 mg fasted); Type 1 tablet - part 2 (2 x 200 mg fed); Type 1 tablet - part 2 (200 mg fasted); Type 1 tablet - part 2 (200 mg fed)
Drug: Padsevonil type 2 Tablet — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Subjects will receive a padsevonil type 2 tablet in a pre-specified sequence during the Treatment Period
  Arms: Type 2 tablet - part 1
Drug: Padsevonil type 3 Tablet — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Subjects will receive a padsevonil type 3 tablet in a pre-specified sequence during the Treatment Period.
  Arms: Type 3 tablet - part 1
Drug: Padsevonil type 4 Tablet — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Subjects will receive a padsevonil type 4 tablet in a pre-specified sequence during the Treatment Period.
  Arms: Type 4 tablet - part 1
Drug: Padsevonil type 5 Tablet — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Subjects will receive a padsevonil type 5 tablet in a pre-specified sequence during the Treatment Period.
  Arms: Type 5 tablet - part 1

SUMMARY:
The purpose of the study in Part 1, is to evaluate (under fasted conditions) the plasma pharmacokinetics (PK) of padsevonil (PSL) using 4 PSL product variants against a PSL reference tablet and in Part 2, to evaluate the PK of PSL using a PSL reference tablet under fed and fasted conditions at 200 mg and 400 mg.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age, inclusive, at the time of signing the informed consent form (ICF)
* Study participants must be overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Study participants must have a body weight of at least 50 kg for males and 45 kg for females and body mass index within the range 18 to 35 kg/m2 (inclusive)
* Study participants who are male or female:

  1. A male participant must agree to use contraception during the treatment period and for at least 7 days after the last dose of study treatment and refrain from donating sperm during this period
  2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

     * Not a woman of childbearing potential (WOCBP) OR
     * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days (or 5 terminal half-lives) after the last dose of study medication

Exclusion Criteria:

* Study participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study or a history of schizophrenia, or other psychotic disorder, bipolar disorder, or severe unipolar depression. The presence of potential psychiatric exclusion criteria will be determined based on the psychiatric history collected at Screening
* Study participant has a history or presence of/significant history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Study participant has a history or present condition of respiratory or cardiovascular disorders, (eg, cardiac insufficiency, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia, or myocardial infarction)
* Study participant has had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Study participant has used hepatic enzyme-inducing drugs (eg, glucocorticoids, phenobarbital, isoniazid, phenytoin, rifampicin, etc) within 2 months prior to the first dose of study medication. In case of uncertainty, the Medical Monitor should be consulted
* Study participant has participated in another study of an investigational study medication (and/or an investigational device) within the previous 60 days before Screening (or 5 half-lives, whichever is longer) or is currently participating in another study of an investigational study medication (and/or an investigational device)
* Study participant has made a blood donation or has had a comparable blood loss (>400 mL) within the last 3 months prior to the Screening Visit or has made plasma donation within last month prior to the Screening Visit
* Study participant smokes more than 5 cigarettes per day (or equivalent) or has done so within 6 months prior to the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
AUC0-t of padsevonil type 1 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 2 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 3 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 4 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 5 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 1 tablets (2x200 mg, fasted) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 1 tablets (2x200 mg, fed) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 1 tablets (200 mg, fasted) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC0-t of padsevonil type 1 tablets (200 mg, fed) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC(0-t): Area under the plasma concentration-time curve from time zero to time t
AUC of padsevonil type 1 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 2 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 3 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 4 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 5 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 1 tablets (400 mg, fasted) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 1 tablets (400 mg, fed) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 1 tablets (200 mg, fasted) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC: Area under the concentration-time curve from time 0 to infinity
AUC of padsevonil type 1 tablets (200 mg, fed) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  AUC: Area under the concentration-time curve from time 0 to infinity
Cmax of padsevonil type 1 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 2 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 3 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 4 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 5 tablets during part 1 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 1.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 1 tablets (400 mg, fasted) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 1 tablets (400 mg, fed) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 1 tablets (200 mg, fasted) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  Cmax: Maximum observed plasma concentration
Cmax of padsevonil type 1 tablets (200 mg, fed) during part 2 | Plasma samples will be taken at: predose and 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8 ,12, 24, 36, 48, 60, and 72 hours during part 2.
  Cmax: Maximum observed plasma concentration

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From Baseline up to Day 35
  An Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Incidence of Serious Adverse Events (SAEs) | From Baseline up to Day 35
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.